CLINICAL TRIAL: NCT01820507
Title: Prevention of Post-extubation Respiratory Failure in High Risk Patients by High-flow Conditioned Oxygen Therapy Versus Standard Oxygen Therapy
Brief Title: Extubation Failure Prevention in High Risk Patients by High-flow Conditioned Oxygen Therapy vs. Standard Oxygen Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment, interim analysis
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Rafael Fernandez, Head of Intensive Care Department, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIC 12/85
Record Dates: First submitted 2013-03-26; First posted 2013-03-28 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Respiratory Failure
Keywords: Post-extubation respiratory failure; Endotracheal intubation; Mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Cannula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Flow Conditioned Oxygen Therapy (Experimental): Intervention: The Optiflow(R) device supplies oxygen in controlled concentrations and at high flow (from 10 to 70 liters/min) through special nasal cannulae. The device also humidifies the gases mixtures up to 100% relative humidity.
  Interventions: Device: Optiflow (Fisher&Paykel)
- Standard Oxygen Therapy (Active Comparator): The standard way of oxygen supply after extubation is either by nasal cannulae at flow between 1 and 5 liters/min or by mask with controlled oxygen concentration from 24% to 50%.
  Interventions: Device: Nasal cannulae or controlled oxygen concentration mask

INTERVENTIONS:
Device: Optiflow (Fisher&Paykel) — The described method of oxygen supply will be maintained continuously for the first 24 hours after extubation.
  Other Names: High Flow Conditioned Oxygen Therapy
  Arms: High Flow Conditioned Oxygen Therapy
Device: Nasal cannulae or controlled oxygen concentration mask — The described method of oxygen supply will be maintained continuously for the first 24 hours after extubation.
  Other Names: Standard Oxygen Therapy
  Arms: Standard Oxygen Therapy

SUMMARY:
Failure of extubation after mechanical ventilation is a frequent and deleterious issue. Main reasons for failure are hypoxemia, secretions retention, lung collapse and excessive work of breathing. Most of this issues can be partly counterbalanced by a device named "High flow conditioned oxygen therapy (HFCO)". Then, our hypothesis is that HFCO may reduce the incidence of respiratory failure after extubation in patients with high risk for failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients mechanically ventilated for > 48 hours and at least one of the following:
* >65 years
* cardiac failure as the primary indication of mechanical ventilation
* Chronic Obstructive Pulmonary Disease
* Severity score (APACHE II >12 points) the extubation day
* Body Mass Index >30
* inability to manage respiratory secretions
* 1 failed spontaneous breathing trial
* 1 comorbidity
* 7 days under mechanical ventilation

Exclusion Criteria:

* <18 years
* tracheotomized patients
* recent facial or cervical trauma/surgery
* active gastro-intestinal bleeding
* lack of cooperation
* patients with any failed spontaneous breathing trial because of hypercapnia development.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Respiratory failure after extubation | 72 hours
  Severe hypoxemia (PaO2/Fraction of inspired O2 < 200), hypercapnia (PaCO2 > 50), respiratory acidosis (arterial pH < 7.30), severe tachypnea (>40x')

SECONDARY OUTCOMES:
Survival | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Fernandez, MD, Principal Investigator — Fundacio Althaia
Locations (1):
- ICU. Fundacio Althaia, Manresa, Barcelona, Spain

REFERENCES:
- [Derived] Fernandez R, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Masclans JR, Lesmes A, Panadero L, Hernandez G. High-flow nasal cannula to prevent postextubation respiratory failure in high-risk non-hypercapnic patients: a randomized multicenter trial. Ann Intensive Care. 2017 Dec;7(1):47. doi: 10.1186/s13613-017-0270-9. Epub 2017 May 2. PMID 28466461